CLINICAL TRIAL: NCT02315118
Title: Pilot Study of Autologous T Lymphocytes With Antibody-Dependent Cell Cytotoxicity in Patients With CD20-Positive B-Cell Malignancies
Brief Title: Pilot Study of Autologous T Lymphocytes With ADCC in Patients With CD20-Positive B-Cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/00584
Record Dates: First submitted 2014-11-27; First posted 2014-12-11 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Rituximab; Interleukin-2; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T-cell therapy + Rituximab + IL-2 (Experimental): Patients will undergo apheresis procedure and T cell expansion will be done in the laboratory. All patients will receive Rituximab on day -2 and IL-2 three times per week for one week starting on day -1 (dose 1 of 3). IL-2 dosing will be continued 3 times per week for one week (3 doses total).
  On Day 0, T cell modification in the laboratory and T cell infusion in the patient will be done.
  A disease status evaluation will be conducted approximately 4 weeks post-T cell infusion.
  Interventions: Drug: T-cell therapy + Rituximab + IL-2

INTERVENTIONS:
Drug: T-cell therapy + Rituximab + IL-2 — * T cells collection
  * T cells expansion and modification in the laboratory
  * T cells infusion back to the patients
  Other Names: T-cell therapy

SUMMARY:
Despite advancement in chemotherapy, radiotherapy and haematopoietic stem cell transplant (HSCT), and the recent introduction of more targeted therapies, a substantial proportion of patients with B-cell malignancies, such as B-cell chronic lymphocytic leukemia (CLL) and B-cell non-Hodgkin's lymphoma (NHL) still succumb to their malignancies. For CLL and low-grade NHL, cure is achievable only with HSCT but such aggressive approach is not justified as the initial therapy for most patients who have indolent disease; when disease has progressed, transplant is either not feasible or ineffective. For high-grade B-cell NHL, the availability of Rituximab has improved disease outcome but treatment failure portends nearly inevitable death from disease or treatment-related complications. Thus, newer, more effective therapies for patients with B-cell malignancies are urgently needed.

The present study translates recent laboratory findings into clinical application. In patients with B-cell malignancies receiving the anti-CD20 antibody Rituximab as standard therapy, the study aims to assess the feasibility and safety, as well as explore the efficacy, of infusing autologous T-lymphocytes engineered to express a CD16-41BB-CD3zeta chimeric receptor which mediates antibody-dependent cell cytotoxicity. Receptor expression is achieved by electroporation of mRNA.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6 months to 80 years old.
2. i) Diagnosis of aggressive CD20+ B-NHL with measurable tumor burden (by imaging, flow cytometry and/or PCR) post-treatment. This includes patients with persistent disease following more than 2 lines of chemotherapy, as well as patients who relapse following autologous transplantation, and in whom further salvage therapy has produced only a partial remission or where no effective salvage therapy available. Patients with bulky disease who require immediate salvage therapy will not be eligible.

   OR ii) Diagnosis of poor risk indolent CD20+ B-NHL or Chronic Lymphocytic Leukemia. This includes high risk CLL cases with early relapse (<12 months following purine analog containing treatment or <24 months following autologous transplant), or with 17p deletion needing treatment, and who are not candidates (or refuses) allogeneic transplantation. Patients with advanced progressive indolent B-NHL with relapsed, refractory disease who have failed more than 2 lines of treatment (including autologous transplantation) may also be considered.
3. Shortening fraction greater than or equal to 25%.
4. Glomerular filtration rate greater than or equal to 50 ml/min/1.73 m2.
5. Pulse oximetry greater than or equal to 92% on room air.
6. Direct bilirubin less than or equal to 3.0 mg/dL (50 mmol/L).
7. Alanine aminotransferase (ALT) is no more than 2 times the upper limit of normal unless determined to be directly due to disease.
8. Aspartate transaminases (AST) is no more than 2 times the upper limit of normal unless determined to be directly due to disease.
9. Karnofsky or Lansky performance score of greater than or equal to 50.
10. No clinical history of or overt autoimmune disease.
11. No past history of previous severe adverse reactions to rituximab, eg. cytokine release syndrome
12. Has recovered from all acute NCI Common Toxicity Criteria grade II-IV non-hematologic acute toxicities resulting from prior therapy per the judgment of the PI.
13. Is not receiving more than the equivalent of prednisone 10 mg daily.
14. Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
15. Not lactating.

Exclusion Criteria:

Failure to meet any of the inclusion criteria

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Performance status assessed by age-dependent Performance Scores | One-month (30 days) after the last T cell infusion
  Using KARNOFSKY PERFORMANCE STATUS SCALE (Recipient Age ≥ 16 years) and LANSKY PERFORMANCE STATUS SCALE (Recipient Age < 16 years)
Toxicity criteria | One-month (30 days) after the last T cell infusion
  Participants will be monitored for toxicity for a period of one-month (30 days) after the last T cell infusion. Monitored toxicities will include the following:
  1. grades III-IV allergic reactions related to infusion;
  2. grade IV neutropenia lasting greater than 28 days;
  3. grade IV infection uncontrolled for greater than 7 days;
  4. grade IV other adverse events;
  5. treatment-related death (grade V).
Disease response criteria | One-month (30 days) after the last T cell infusion and at intervals thereafter till progression (approximately every 3 months for about a year)
  Response criteria follow those defined by NCCN Guidelines version 4.2011 for CLL and NHL.
  For monitoring of treatment response, patients with CLL and NHL will have PET-CT scan at approximately 1 month before and after infusion and at intervals thereafter till progression. Peripheral blood and bone marrow studies (the latter only if bone marrow is involved pre-treatment) will be done to determine levels of residual disease by using established flow cytometric and molecular MRD assays.
Persistence of CD16+ T cells and impact on B cell function | Up to approximately month
  1. The in vivo expression of anti-CD16V-BB-zeta on T cells will be monitored by flow cytometry. For this purpose, 10 ml of blood will be taken on Days 0, 1 and every other day after each infusion until infused T cells expressing the receptor become undetectable.
  2. Longer term impact on the suppression of B cell function will also be monitored by assaying B cell numbers and immunoglobulin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Poon, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore; Yeh Ching Linn, MBBS, MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Kudo K, Imai C, Lorenzini P, Kamiya T, Kono K, Davidoff AM, Chng WJ, Campana D. T lymphocytes expressing a CD16 signaling receptor exert antibody-dependent cancer cell killing. Cancer Res. 2014 Jan 1;74(1):93-103. doi: 10.1158/0008-5472.CAN-13-1365. Epub 2013 Nov 6. PMID 24197131